CLINICAL TRIAL: NCT04625543
Title: Neoadjuvant Immunotherapy Combined With Neoadjuvant Chemotherapy for Locally Advanced Esophageal Cancer: an Open Label, Randomized Control, Phase II Trial
Brief Title: Neoadjuvant Immunotherapy to ESCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient money
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Sang Shaowei, Associate Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO-PD-1-II-ESCC
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Esophagus SCC
Keywords: ESCC; PD-1/PD-L1; Randomized controlled clinical trial; neoadjuvant
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Paclitaxel; Cisplatin; TP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Neoadjuvant immunotherapy (PD-1) plus concurrent chemotherapy (paclitaxel + Cisplatin) will be applied to patients with locally advanced esophageal squamous cell carcinoma with PD-L1>=10% before surgery.
  Interventions: Drug: Sintilimab Injection plus Paclitaxel and Cisplatin
- controll group (Active Comparator): Neoadjuvant chemotherapy (paclitaxel + Cisplatin) will be applied to patients with locally advanced esophageal squamous cell carcinoma with PD-L1>=10% before surgery.
  Interventions: Drug: Paclitaxel and Cisplatin

INTERVENTIONS:
Drug: Sintilimab Injection plus Paclitaxel and Cisplatin — Paclitaxel 150mg/m2 on day 1, every 3 weeks, for two cycles; Cisplatin 70mg/m2 on day 1, every 3 weeks, for two cycles; Sintilimab Injection 200mg on day 22; 4-6 weeks after completion of preoperative therapy, Mckeown esophagectomy will be performed if there is no contraindication.
  Arms: intervention group
Drug: Paclitaxel and Cisplatin — Paclitaxel 150mg/m2 on day 1, every 3 weeks, for two cycles; Cisplatin 70mg/m2 on day 1, every 3 weeks, for two cycles; 4-6 weeks after completion of preoperative therapy, Mckeown esophagectomy will be performed if there is no contraindication.
  Arms: controll group

SUMMARY:
Currently, surgery after neoadjuvant chemoradiotherapy is the standard treatment for patients with locally advanced esophageal cancer, but the recurrence rate is high and the 5-year survival rate is low. Immunotherapy shows a potential treatment for esophageal cancer. Immunocheckpoint (PD-1/PD-L1) inhibitors can activate tumor immunity. The guidelines have recommended it as a sencond-line therapy. However, there is still lack of the evidence for its efficacy as a neoadjuvant therapy. This study is to conduct a randomized controlled, open label, phase II clinical trial to evaluate the efficacy and safety of neoadjuvant immnotherapy combined with neoadjuvant chemotherapy for locally advanced esophageal squamous cell carcinoma (ESCC) patient with PD-L1 (CPS>=10%) positive.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participated and sign information consent;
2. Age 18-70, male or female;
3. Locally advanced esophageal cancer diagnosed by pathology, Clinical tumor stage should be II-IVa; tumor located at the lower middle segment;
4. No previous chemoradiotherapy or immunotherapy;
5. PD-L1 expression >=10%;
6. Have a performance status of 0 or 1 on the ECOG Performance Scale;
7. Demonstrate adequate organ function as defined below (excluding the use of any blood components and cytokines during the screening period): Absolute neutrophil count (ANC) ≥1.5*109 /L; Platelet ≥100*109/L; Hemoglobin ≥ 9 g/dL; Serum albumin≥3g/dL; Bilirubin≤1.5 x ULN; ALT and AST≤2.5 ULN; Serum creatinine ≤1.5 x ULN or creatinine clearance ≥40mL/min; LVEF>=50%; Urine protein<++; INR<1.5 and APTT<1.5;
8. Female subject must have taken reliable contraceptive measures of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. and be willing to use an appropriate method of contraception during the trial and 8 weeks after the last administration of the test drug. Male subject should agree to use appropriate contraceptive methods or to have been surgically sterilized during the trial and 8 weeks after the last administration of the test drug.

Exclusion Criteria:

1. Any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitritis, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction);
2. Asthma requiring medical intervention with bronchodilators was not included.
3. Subjects with history of severe allergy;
4. There are clinical symptoms or diseases of the heart that are not well controlled, such as: heart failure above grade 2 by the Criteria of NYHA; unstable angina pectoris; myocardial infarction occurred within 1 year; Clinically meaningful supraventricular or ventricular arrhythmias require treatment or intervention;
5. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), or has known active Hepatitis B (e.g. HBV DNA≥ 2000IU/ml or copy number ≥104/ml;) or Hepatitis C (e.g. HCV antibody positive);
6. Systematic glucocorticoid therapy is administered one week prior to neoadjuvant therapy;
7. Subjects who are participating other drug clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rate | 30 days after the second cycle of treatment(each cycle is 21 days)
  MPR is defined as 10% or fewer viable cancer cells in the hematoxylin and eosin (H&E)-stained slides from the resected tumor following neoadjuvant treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | at the end of the second cycle of treatment(each cycle is 21 days)
  ORR determines the tumor shrinkage rate, tumor boundary and the adhesion of tumor
2-year progression-free survival (PFS) | every 3 months (up to 24 months)
  From date of surgery until the date of first documented progression or date of death from any cause
The incidence of adverse events | the day from the first treatment cycle
  Safety will be evaluated for all treated patients using CTCAE V 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shaowei Sang, Doctor, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China